CLINICAL TRIAL: NCT00233506
Title: A Dose-Finding Study of CpG 7909 in Previously Treated Chronic Lymphocytic Leukemia
Brief Title: A Dose Finding Study of CpG in Patients With Chronic Lymphocytic Leukemia Who Have Been Previously Treated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Mayo Clinic (Other); Pfizer (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Link, Brian K, Professor, University of Iowa
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200402002
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CpG 7909; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ProMune

ARMS (2):
- CPG 7909 IV (Experimental): Intravenous infusions will be administered with a standard infusion pump beginning at 125 cc/hr through an intravenous catheter (central or peripheral).
  Interventions: Drug: CpG 7909
- CPG 7909 SQ (Experimental): Subcutaneous injections should be administered in the abdominal wall, upper arm, hip, or anterior thigh. If the volume of injection exceeds 1.5 ml, the volume should be divided into equal injections at a volume less than 1.5 ml and administered in different areas of the body. The maximum dose level on this trial may require 5 - 6 injections at an equal number of sites.
  Interventions: Drug: CpG 7909

INTERVENTIONS:
Drug: CpG 7909

SUMMARY:
* CpG has the potential to stimulate the immune system
* this study will evaluate the safety of CpG given sub-q or IV
* purpose is to measure biological changes in CLL cells after receiving CpG

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL
* CLL previously treated
* Hemoglobin >/= 10
* Platelets >/= 50,000
* Neutrophils >= 1,000 -

Exclusion Criteria:

* patients with brain mets
* patients with autoimmune disease
* patients on corticosteroids or immunosuppressants
* patients with uncontrolled intercurrent illness
* pregnant women
* HIV patients receiving combination anti-retroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2004-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | at study completion

SECONDARY OUTCOMES:
response | at end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Brian Link, MD, Principal Investigator — UIHC; Clive Zent, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Mayo Clinic, Rochester, Minnesota